CLINICAL TRIAL: NCT01673139
Title: Effect of 3 Years of Exercise in Patients With Atrial Fibrillation - A Generation 100 Substudy
Brief Title: Effect of 3 Years of Exercise in Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); SINTEF Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012/978b
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Exercise
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate exercise (Experimental): Moderate exercise
  Interventions: Behavioral: Moderate exercise
- Control (Experimental): Control group
  Interventions: Behavioral: Control
- Interval exercise (Experimental): interval exercise
  Interventions: Behavioral: Interval exercise

INTERVENTIONS:
Behavioral: Interval exercise — 4 times of 4 minutes intervals at an intensity of 90-95% of maximum heart rate and active pauses of 3 minutes between intervals. 3 times a week for 3 years.
  Arms: Interval exercise
Behavioral: Moderate exercise — Moderate exercise with pulse about 70% of max pulse; 3 times a week for 3 years.
  Arms: Moderate exercise
Behavioral: Control — Given information on recommendations for physical activity.
  Arms: Control

SUMMARY:
This is a substudy of "Generation 100". The investigators will follow the persons with atrial fibrillation to see if 3 years of interval or moderate exercise affects the burden of atrial fibrillation, symptoms, use of health services or echocardiographic findings.

ELIGIBILITY:
Inclusion Criteria:

* Included in the "Generation 100 study"
* Atrial fibrillation diagnosis verified by ECG

Exclusion Criteria:

-

Ages: 70 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in burden of atrial fibrillation | At baseline and 3 years
  Burden of atrial fibrillation; measured by Holter monitor and the patient.

SECONDARY OUTCOMES:
Size of left ventricle | At baseline and 3 years
  Echocardiographic measures
Quality of life | At baseline and 3 years
  Measured with SF-36
Endothelial function | At baseline and 3 years
  Diameter of brachial artery measured by ultrasound.
Maximal oxygen uptake | At baseline and 3 years
Atrial extrasystoles | At baseline and 3 years
  Measured with Holter monitor
Number of hospitalisations with atrial fibrillation as main diagnosis | Total number during the 3 year intervention period
Total number of electrical cardioversions | During the 3 years of intervention
  Number of electrical cardioversions because og atrial fibrillation
Change in burden of atrial fibrillation | Baseline and 1 year
  Measured by Holter and the patient.
Size of left atrium | Baseline and 1 year
  Echocardiography
Function of left atrium | At baseline and 3 years
  Echocardiographic measures
Function of left ventricle | At baseline and 3 years
  Echocardiographic measures
Size of left atrium | At baseline and 3 years
  Echocardiographic measures
Symptom burden | At baseline and 3 years
  Measured with Symptom and Severity Checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paal Loennechen, PhD, Study Chair — St. Olavs Hospital
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway